CLINICAL TRIAL: NCT06790550
Title: Examination of Music's Demonstration to Self-Injection, Fear of Testing and Pain in Patients With Type 2 Diabetes
Brief Title: Music Effect on the Self-Injection, Testing Fear and Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Hamdiye ARDA SÜRÜCÜ, PROFESSOR, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DICLE-ARDASURUCU-002
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Insulin; Fear; Pain; Injection; Music Therapy
Keywords: type 2 diabetes mellitus; Insulin; fear; pain; insulin injection; music
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Pain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: study group and control group
Who Masked: Participant
Masking Description: They do not know the experimental or control procedures that take place
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): Music will be played during the insulin injection process
  Interventions: Other: Music Therapy
- Control group (Music free) (No Intervention): patients without of experimental Music

INTERVENTIONS:
Other: Music Therapy — Music will be played during the insulin injection process
  Arms: Music group

SUMMARY:
Diabetes is a chronic and broad-spectrum metabolic disorder characterized by hyperglycemia that occurs due to relative or absolute insulin deficiency or "insulin resistance" developed against insulin action in peripheral tissues, affecting many organs and causing multisystem involvement. Metabolic function continues to deteriorate after diagnosis, leading to worsening glycemic control and insulin therapy becoming necessary. However, patients may have difficulty adhering to insulin therapy. Fears about injections are common in both adults and children and, as research shows, are a major reason why people with diabetes avoid taking insulin. Addressing these fears is an important part of helping patients reduce their risk of diabetes-related complications. Helping patients manage their replacement pain may help reduce the effects of needle fear in the future. There are a number of strategies that can ease the pain.The use of music in pain management has advantages such as being reliable, cheap, and having no side effects, as well as reducing postoperative pain reports. Music distracts the individual from negative stimuli and allows them to focus on something they enjoy, thus reducing pain and anxiety. Music therapy has also been shown to have sedative-protective effects and reduce stress hormone levels. Listening to preferred music can distract and reduce the pain and negative emotions associated with an unpleasant experience.

DETAILED DESCRIPTION:
Research Type:

The research will be conducted as a randomized controlled experimental model.

Research Universe and Sample:

The research sample will consist of patients diagnosed with Type 2 Diabetes hospitalized in a State Hospital. The sample of the research is expected to consist of 100 volunteer Type 2 Diabetes patients who applied to the State Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least one year
* Self-administering insulin injection
* Self-administering glucometer, insulin pen or insulin pump

Exclusion Criteria:

* poor mental health
* Having gestational diabetes mellitus or Type 1 diabetes
* no hearing problems

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Before insulin administration on day, Time Frame: After two insulin administration on the second day
  The scale is used to assess subjectively perceived pain. It is a 10 cm (100 mm) ruler with no pain on one end and the "most severe pain" on the other. The individuals participating in the study are asked to mark the intensity of pain they are currently feeling, explaining that the number "0" on the scale means "I feel no pain" and that the intensity of pain increases as the numbers increase, and the number "10" means "I feel the most severe pain". An increase in the score obtained from the scale in the assessment indicates that the pain is increasing. Each patient will be administrated three times.

SECONDARY OUTCOMES:
Diabetes Fear of Self Injecting and Self-testing Questionnaire | Before insulin administrated on day one, Time Frame: After two insulin administration on the second day.
  Questionnaire measures fear of self-injection and testing in diabetic individuals who require insulin. Questionnaire, which contains 15 statements, consists of two sub-dimensions: fear of self-injecting (6 statements) and fear of self-testing (9 statements). Each statement has a four-point Likert-type scoring ranging from 0 to 3 (0= almost never, 1= sometimes, 2= often, 3= almost always). The evaluation of the questionnaire form can be done by taking the average or raw score for the two sub-dimensions and the entire form. When taken as raw score, self-injection fear score varies between 0-18, self-testing fear score between 0-27, and total fear score between 0-45. Increasing score indicates increasing fear. Each patient will be administrated three times.

CONTACTS AND LOCATIONS:
Locations (1):
- Dicle Univertsity, Diyarbakır, South East, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No